CLINICAL TRIAL: NCT00685737
Title: A Randomized Placebo Controlled Double Blind Two Period Cross-Over Study to Assess the Safety and Pharmacokinetics and Pharmacodynamics of Oral Dosages of 1-MNA, (A Hypolipidemic Agent) in Healthy Volunteers
Brief Title: Safety of a Hypolipidemic Agent in Healthy Normal Volunteers
Acronym: PNAI-002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmena North America (Industry)
Responsible Party: Charles Ballow, Pharm D. FACCP, Buffalo Clinical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PNAI-002
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 1-MNA-Low Dose
  Interventions: Drug: 1-MNA
- 2 (Active Comparator): 1-MNA-High Dose
  Interventions: Drug: 1-MNA
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1-MNA — Capsule
  Arms: 1; 2
Drug: Placebo — Capsule
  Other Names: Placebo Comparator
  Arms: 3

SUMMARY:
The Purpose of this study is to determine the safety and tolerability of 1-MNA, a drug that is intended to be used in the treatment of elevated levels of blood fats. This study will determine the way that 1-MNA is handled by the body, and will also determine its effect on commonly measured blood fat parameters.

DETAILED DESCRIPTION:
Dyslipidemia is a major risk factor for coronary artery disease (CAD) and its management is important in preventing the occurrence of cardiovascular events. Dyslipidemia occurs when there is an imbalance in the metabolism and clearance of lipoproteins resulting in lipoprotein overproduction or deficiency. Lipid related risk factors for atherosclerotic coronary artery disease include elevated levels of total cholesterol (TC), triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), intermediate-density lipoprotein cholesterol (IDL-C), very low-density lipoprotein cholesterol (VLDL-C) and reduced concentrations of high-density lipoprotein cholesterol (HDL-C). This lipid risk profile frequently occurs in association with other cardiovascular risk factors (e.g., obesity, elevated blood pressure, diabetes mellitus), and is associated with premature atherosclerosis (NCEP, 2002).

The Main purpose of this study is to formally evaluate the safety and pharmacokinetics and pharmacodynamics of 1-MNA, a hypolipidemic agent with previous human exposure in normal subjects and patients with Hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Good health (based on medical history, physical examination, electrocardiogram, and clinical laboratory tests)
* Non-smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the Screening visit)
* Between 18 and 50 years old (inclusive)
* Body weight within 20% of the desirable weight for adults at the Screening visit
* Able to execute informed written consent (informed consent must be obtained for all subjects before enrollment in the study.
* Willingness to abstain from alcohol and xanthine-containing food and beverages for the duration of each treatment period
* Willingness to remain in the clinic for the inpatient portions of the study
* Female subjects must be non-pregnant and either surgically sterile, postmenopausal for a least 1 year, or using an acceptable method of contraception defined as an oral, implanted, or transdermal contraceptive plus one of the following barrier methods: diaphragm with spermicidal cream/jelly or use of a condom by sexual partner.

Exclusion Criteria:

* Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years
* Unwilling or unable to comply with the protocol or reside in the study unit during the study period or to cooperate fully with the principal investigator and site personnel
* Has used any 1) prescription medication within 14 days prior to treatment in either treatment period or 2), or any over-the-counter (OTC) medication, herbal preparations, and/or vitamins within 48 hours prior to the start of study MNA administration on either treatment period of this study.
* Has a clinically abnormal ECG
* Has a serum potassium, sodium, calcium, or magnesium level that is not within normal limits or has other vital signs or clinical laboratory values at the screening visit that are deemed by the principal investigator to make the subject an inappropriate candidate for the study
* Has taken any other investigational drug during the 30 days prior to screening visit
* Has donated or lost more than a unit of blood within 30 days prior to screening visit
* History of renal, hepatic, gastrointestinal, cardiovascular, or hematologic disease
* Serious mental or physical illness within the past year
* Has any condition(s) that in the investigator's opinion would: a) warrant exclusion from the study or b) prevent the subject from completing the study
* Have a positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody at screening
* Be a female subject with a positive serum pregnancy test or who is breast-feeding at screening
* Be unable to understand verbal and/or written English or any other language in which a certified translation of the informed consent is available
* Has a history of hypersensitivity or allergic reaction to Niacin or Nicotinamide
* Has had prior exposure to MNA
* Has a Mental capacity that is limited to the extent that the subject cannot provide legal consent or understand information regarding the side effects or tolerance of the study drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The single dose pharmacokinetics and safety of 1-MNA and an assessment of any gender-based differences in plasma pharmacokinetics | Over 24 hours following a dose

SECONDARY OUTCOMES:
The effect of 1-MNA on triglycerides and lipase activity and lipid profiles after single oral dosages | Over 24 hours following a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Ballow, Pharm D., Principal Investigator — Buffalo Clinical Research Center
Locations (1):
- Buffalo Clinical Research Center, Buffalo, New York, United States